CLINICAL TRIAL: NCT03082196
Title: Phase 2 Efficacy Evaluation Of Advantage Anti-Caries Varnish
Brief Title: Efficacy Of A PVP-I Fluoride Varnish
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advantage Dental Services, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2016-12-02
Record Dates: First submitted 2017-03-13; First posted 2017-03-17 (Actual); Results first posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Dental Caries
Keywords: sodium fluoride; povidone iodine; varnish
MeSH Terms: conditions — Dental Caries | interventions — Bifluorid 12

STUDY DESIGN:
Intervention Model Description: Single-center, double-blind, controlled Phase 2 study with parallel groups of children.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study personnel except for designated personnel in the data center will be blinded to the participant treatment assignment. In order to maintain blinding, the caries scoring examinations will precede the application of test varnishes at baseline. The staff member applying these varnishes will not perform the caries scoring exams in order to eliminate examiner bias and ensure blinding to treatment assignment. Test drug and comparator are packaged identically.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test varnish (Experimental): Advantage Anti-Caries Varnish. The active ingredients are Povidone Iodine and Sodium Fluoride .
  Interventions: Drug: Test varnish
- Standard varnish (Active Comparator): The active control varnish will be the same fluoride varnish without iodine with an appropriate FDA approved food dye added to match the color of the test agent. There will be no difference in the treatment and control varnishes except for the povidone iodine.
  Interventions: Drug: Standard varnish

INTERVENTIONS:
Drug: Test varnish — Topical application of test varnish to the teeth 4 times per year.
  Arms: Test varnish
Drug: Standard varnish — Topical application of test varnish to the teeth 4 times per year
  Other Names: sodium fluoride varnish
  Arms: Standard varnish

SUMMARY:
The purpose of the study is to determine the efficacy of Advantage Anti-Caries Varnish. Single-center, double-blind, controlled Phase 2 study with parallel groups of children. Subjects will be stratified by early childhood education center and then randomized to receive either test varnish or control varnish topically to the teeth. Treatment will be administered quarterly for up to 24 months. The primary outcome is surface-level primary molar caries increment (d2-4mfs) at 24- months post baseline.

DETAILED DESCRIPTION:
Objectives:

Primary

- To determine if Advantage Anti-Caries Varnish (test varnish) is superior to a control varnish containing only fluoride in the prevention of new caries lesions.

Secondary

* To establish that the response of child participants to the test varnish was not inferior to the control varnish

ELIGIBILITY:
Inclusion Criteria:

1. The subject's parent or legal guardian must provide signed and dated informed consent (parent permission form).
2. The subject's parent or legal guardian of the subject must be willing and able to comply with study requirements.
3. The subject is aged 60-84 months at the time of enrollment.
4. The subject must be in good general health as evidenced by parent report.

Exclusion Criteria:

1. Known allergy to iodine
2. Known allergy to seafood
3. Known hypersensitivity to fluoride varnish
4. Diagnosis of thyroid disease
5. Chronic, prophylactic use of antibiotics
6. Treatment with another investigational drug or other intervention within 30 days preceding the Baseline Visit.

Ages: 60 Months to 84 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 284 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Milgrom, DDS, Study Chair — Advantage Silver Dental Arrest, LLC
Locations (1):
- Pohnpei State Hospital, Kolonia, Pohnpei State, Micronesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Milgrom P, Tut O, Rothen M, Mancl L, Gallen M, Tanzer JM. Addition of Povidone-Iodine to Fluoride Varnish for Dental Caries: A Randomized Clinical Trial. JDR Clin Trans Res. 2021 Apr;6(2):195-204. doi: 10.1177/2380084420922968. Epub 2020 May 21. PMID 32437626
- [Derived] Milgrom P, Tut O, Rothen M, Mancl L, Gallen M, Tanzer JM. Efficacy evaluation of an anti-caries varnish: protocol for a phase II randomised controlled trial. BMJ Open. 2017 Jun 30;7(6):e017866. doi: 10.1136/bmjopen-2017-017866. PMID 28667230

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Varnish | Standard Varnish
Started | 142 | 142
Completed | 133 | 129
Not Completed | 9 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Varnish | Standard Varnish | Total
Number analyzed (Participants) | 142 | 142 | 284
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 142 | 142 | 284
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 64 | 140
  Male | 66 | 78 | 144
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 142 | 142 | 284
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 142 | 142 | 284
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Micronesia | 142 | 142 | 284

OUTCOME MEASURES:

1. Primary Outcome: Dental Caries for Primary Molars Sound at Baseline
Description: The primary outcome will be the surface-level primary molar caries increment (d2-4mfs) at two years post baseline. Caries, as measured by d2-4mfs, is the total number of surfaces with decay into the enamel (2), dentin (3) or pulp (4), missing due to caries (m), or filled with amalgam, composite or other filling material (f). This scale records whether caries is detected in any of the 5 surfaces of the tooth for up to 8 primary molar teeth that were sound at baseline, and has a range of 0 to 40. Higher values indicate a greater number of caries.
Time Frame: 24 months
Population: The analysis population is based on the 139 participants with sound molars and baseline and follow-up at 24-months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Varnish | Standard Varnish
Number analyzed (Participants) | 72 | 67
units on a scale | 2.3 (2.8) | 3.3 (2.7)
Statistical Analysis 1: Comparison: Test Varnish vs Standard Varnish; Test type: Superiority; p = 0.037, t-test, 2 sided; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-1.9 to -0.1] — The direction of the comparison (difference) is the test varnish to the standard varnish. A negative value for the difference indicates a lower caries increment in the test varnish as compared to the standard varnish

2. Primary Outcome: Dental Caries for All Primary Teeth Sound at Baseline
Description: The outcome will be the surface-level primary tooth caries increment (d2-4mfs) at two years post baseline that were sound at baseline. Caries, as measured by d2-4mfs, is the total number of surfaces with decay into the enamel (2), dentin (3) or pulp (4), missing due to caries (m), or filled with amalgam, composite or other filling material (f). This scale records whether caries is detected in any of the 4 or 5 surfaces of the tooth for up to 20 primary teeth that were sound at baseline, and has a range of 0 to 88. Higher values indicate a greater number of caries.
  The measure records whether caries is present on any of the 5 surfaces of the primary molars or 4 surfaces of the other teeth.
Time Frame: 24 months
Population: The analysis population is based on participants with sound primary teeth at baseline and follow-up at 24 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Varnish | Standard Varnish
Number analyzed (Participants) | 126 | 116
units on a scale | 2.0 (2.8) | 2.7 (3.3)
Statistical Analysis 1: Comparison: Test Varnish vs Standard Varnish; Test type: Superiority; p = 0.062, t-test, 2 sided; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.5 to 0.1] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Child Response to First Treatment
Description: Facial Images Scale which measures the child's response using a series of five happy/sad faces from a very unhappy face (5) to a very happy face (1). The minimum value is 1 which corresponds to a very happy face and the maximum value is 5 which corresponds to a very unhappy face. The possible values of the scale are 1, 2, 3, 4, or 5.
Time Frame: After first treatment visit
Population: The analysis population is based on participants who received the first varnish application and completed the Facial Image Scale.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Varnish | Standard Varnish
Number analyzed (Participants) | 141 | 142
units on a scale | 2.3 (1.2) | 2.5 (1.3)
Statistical Analysis 1: Comparison: Test Varnish vs Standard Varnish; Test type: Superiority; p = 0.11, t-test, 2 sided; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to 0.1] — The direction of the comparison (difference) is the test varnish to the standard varnish. A negative value for the difference indicates a "happier" response in the test varnish as compared to the standard varnish

4. Secondary Outcome: Child Response to Fifth Treatment
Description: as for outcome 3
Time Frame: After fifth treatment visit
Population: Analysis population based on participants who received the fifth varnish application and completed the Facial Image Scale.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Varnish | Standard Varnish
Number analyzed (Participants) | 135 | 137
units on a scale | 2.2 (1.1) | 2.1 (1.2)
Statistical Analysis 1: Comparison: Test Varnish vs Standard Varnish; Test type: Superiority; p = 0.74, t-test, 2 sided; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.2 to 0.3] — The direction of the comparison (difference) is the test varnish to the standard varnish. A positive value for the difference indicates an "unhappier" response in the test varnish as compared to the standard varnish

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Test Varnish | Standard Varnish
All-Cause Mortality (participants affected / at risk) | 0/142 | 0/142
Serious Adverse Events (participants affected / at risk) | 3/142 | 2/142
Other Adverse Events (participants affected / at risk) | 43/142 | 49/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Varnish (N=142) | Standard Varnish (N=142)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
fracture, arm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Swelling, pain in knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
tonsilitis (Infections and infestations) | 1 (1) | 0 (0)
rheumatic heart disease (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Varnish (N=142) | Standard Varnish (N=142)
Flu (Infections and infestations) | 30 (35) | 27 (33)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 11 (11)
Cough & fever (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT03082196/Prot_SAP_000.pdf